CLINICAL TRIAL: NCT03098771
Title: Peripheral Blood Autologous CD34+ Cell Transplantation Promotes Angiogenesis in Elderly Patients With Atherosclerotic Ischemia: Study Protocol for a Prospective, Single-center, Open-label, Randomized, Controlled, Clinical Trial
Brief Title: Peripheral Blood Autologous CD34+ Cell Transplantation Promotes Angiogenesis With Atherosclerotic Ischemia for Elderly
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qingdao University (Other)
Responsible Party: Principal Investigator, Lili Xu, Principal Investigator, Qingdao University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QingdaoU_001
Record Dates: First submitted 2017-03-22; First posted 2017-04-04 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Atherosclerotic Ischemic Disease

STUDY DESIGN:
Intervention Model Description: Inpatients of the Qingdao No. 9 People's Hospital will be recruited. Potential participants can contact the project manager via telephone. After providing informed consent, these potential participants will be screened using the inclusion and exclusion criteria.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the cell transplantation group (Experimental): Patients with atherosclerotic lower limb ischemia will be randomly assigned to the cell transplantation group, which peripheral blood CD34+ cells transfected with ActiveMax® recombinant human vascular endothelial growth factor 165 (VEGF165) gene will be transplanted into the muscles of ischemic limbs in elderly patients with atherosclerotic lower limb ischemia.
  Interventions: Procedure: the cell transplantation group
- the control group (Experimental): Patients with atherosclerotic lower limb ischemia will be randomly assigned to the control group, which 9% physiological saline will be injected into the muscles of ischemic limbs.
  Interventions: Drug: the control group

INTERVENTIONS:
Procedure: the cell transplantation group — Patients with atherosclerotic lower limb ischemia will be randomly assigned to the cell transplantation group, which peripheral blood CD34+ cells transfected with ActiveMax® recombinant human vascular endothelial growth factor 165 (VEGF165) gene will be transplanted into the muscles of ischemic limbs in elderly patients with atherosclerotic lower limb ischemia.
  Arms: the cell transplantation group
Drug: the control group — Patients with atherosclerotic lower limb ischemia will be randomly assigned to the control group, which 9% physiological saline will be injected into the muscles of ischemic limbs.
  Other Names: the physiological saline group
  Arms: the control group

SUMMARY:
To verify angiogenesis in elderly patients with atherosclerotic ischemia after peripheral blood autologous CD34+ cell transplantation.

DETAILED DESCRIPTION:
History and current related studies Arteriosclerosis obliterans is a kind of arterial lumen stenosis and occlusive disease, which is caused by the continuous expansion of arterial atherosclerosis and secondary thrombosis. Clinical manifestations are local skin temperature reduction, intermittent claudication, rest pain, ulcers difficult to heal, and gangrene infection.Some patients require amputation or even it is life-threatening. Arteriosclerosis obliterans of lower limbs are commonly treated by surgical treatment, endovascular treatment and non-surgical treatment, but the effect is not very satisfactory.

For the treatment of arteriosclerosis obliterans, stem cell transplantation has achieved great progress in angiogenesis and collateral circulation. There are two main mechanisms of stem cells involved in angiogenesis: (1) Promoting differentiation and maturation of new blood vessels by homing and integration in the damaged vascular plexus; (2) Promoting angiogenesis in ischemic tissue by paracrine of vascular endothelial growth factor (VEGF).In recent years, because of the discovery of endothelial progenitor cells in peripheral blood, the concept of angiogenesis has been renewed. Transplantation of endothelial progenitor cells and bone marrow cells for angiogenesis has become the focus of research. Endothelial progenitor cell and bone marrow cell transplantation have been used to promote angiogenesis in ischemic tissue in order to treat limb ischemia.

Bone marrow stem cell mobilization is used to promote the replication of bone marrow stem cells, so as to increase the number of endothelial progenitor cells in peripheral blood, i.e., the number of stem cells homing to ischemic tissue, and finally accelerating the speed and magnitude of angiogenesis. Fujisaki et al. have confirmed that bone marrow cell mobilizers can significantly stimulate bone marrow hematopoiesis and increase the number of peripheral blood stem cells.Bone marrow cell mobilizer-recombinant human granulocyte colony stimulating factor (rhG-CSF) are used to mobilize bone marrow stem cells to peripheral blood, and to increase the number of peripheral blood stem cells, especially endothelial progenitor cells, so as to treat ischemic diseases using transplanted autologous stem cells, which is called autologous stem cell transplantation. Nevertheless, in animal and human experiments, the proliferation potential and influencing factors of mobilized bone marrow stem cells and peripheral blood endothelial progenitor cells in ischemic tissue require further investigations.

Autologous stem cell transplantation is to transplant stem cells in muscles of ischemic limb, so that new capillaries improve and restore lower limb blood flow, aiming to treat lower limb ischemia. Endothelial progenitor cells and hematopoietic stem cells are thought to come from a common ancestor, and called blood vessel stem cells. They express immature stem cell markers CD34 and CD133. Endothelial progenitor cells migrated from bone marrow to peripheral blood will gradually lose CD133, and the disappearance of CD34 is relatively slow. A large number of basic and clinical studies have confirmed that the transplantation of CD34+ cells can promote angiogenesis in ischemic limbs of experimental animals (partial patients).

Adverse events

1. To record adverse events, including fever, infection, lower limb pain and ulcers, during follow-up at out-patient clinic.
2. If severe adverse events occur, investigators will report details, including the date of occurrence and measures taken to treat the adverse events, to the principle investigator and the institutional review board within 24 hours.

Data collection, management, analysis, open access

1. Data collection: Case report forms will be collected and processed using Epidata software (Epidata Association, Odense, Denmark), collated, and then recorded electronically using a double-data entry strategy.
2. Data management: The locked electronic database will be accessible and locked only by the project manager. This arrangement will not be altered. The Qingdao No. 9 People's Hospital, China will preserve all of the data regarding this trial.
3. Data analysis: A professional statistician will statistically analyze the electronic database and will create an outcome analysis report that will be submitted to the lead researchers. An independent data monitoring committee will supervise and manage the trial data, ensuring a scientific and stringent trial that yields accurate and complete data.
4. Data open access: Anonymized trial data will be published at www.figshare.com.

Statistical analysis

1. Statistical analysis will be performed using SPSS 19.0 software (IBM, Armonk, NY, USA) and will follow the intention-to-treat principle.
2. Normally distributed measurement data will be expressed as means, standard deviation, minimums and maximums. Non-normally distributed measurement data will be expressed as the lower quartile (q1), median and upper quartiles (q3). Count data will be expressed as a percentage.
3. Kolmogorov-Smirnov test will be used to determine normality of measurement data. If data obey the normal distribution, ABI, number of microvessels in the lower limb muscles and number of VEGF-immunoreactive cells will be compared with two-sample t-test between the two groups. Intragroup difference of above indicators will be compared using paired t-test before and 6 months after transplantation. If data do not obey the normal distribution, intergroup and intragroup data will be compared using Mann Whitney U test and Wilcoxon signed-rank test. The incidence of adverse reactions will be compared with Fisher's exact probability test between the two groups 6 months after transplantation.
4. The significance level will be α = 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Elderly patients with arteriosclerosis obliterans (Rutherford classification of class 5: slight tissue defect; class 6: tissue ulceration, gangrene)
* Diabetic foot, Wagnar classification of class 315: deep ulcer, often affecting bone tissue, with deep abscess or osteomyelitis
* Age range: 50-60 years
* Irrespective of gender
* Unilateral limb lesions
* Total occlusion of main blood vessels
* No outflow tract in distal arteries
* Cannot perform open surgery and endovascular surgery
* Signed informed consent

Exclusion Criteria:

* Moderate to severe liver and kidney dysfunction
* Malignant tumor
* Hematological system diseases
* Rheumatic immune system diseases
* Poor stimulating effect on colony stimulating factor
* Thromboangiitis obliterans
* Severe hyperthyroidism
* Endocrine and metabolic diseases such as severe hypothyroidism

Ages: 50 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
ankle-brachial index (ABI) | Change from baseline ankle-brachial index (ABI) at 6 months
  To assess lower limb ischemia. Ankle-brachial index (ABI) is the ratio of the blood pressure at the ankle to the blood pressure in the upper arm (brachium; Appendix 1). The range of ABI of normal persons at resting is between 0.9 and 1.3. Abnormal results: less than 0.8 represents moderate disease; less than 0.5 represents severe disease. The ABI of intermittent claudication patients is mainly between 0.35 and 0.9. The ABI of rest pain patients is often less than 0.4, and the patient will be at risk of amputation. ABI of more than 1.3 indicates vascular wall calcification and loss of vascular contraction.

SECONDARY OUTCOMES:
Number of microvessels in the lower limb muscles | Change from baseline ankle-brachial index (ABI) at 6 months
  To observe the changes in microvessel number.Five fields will be randomly selected under a high power microscope (× 400). High number of microvessels indicates the generation of more new blood vessels.

CONTACTS AND LOCATIONS:
Overall Officials: Lili Xu, Ph.D, Principal Investigator — The Affiliated Hospital of Qingdao University

IPD SHARING:
Plan to Share IPD: Undecided